CLINICAL TRIAL: NCT06684405
Title: Fluoridated Milk is Effective in Prevention of Enamel Caries in Adolescents
Brief Title: Fluoridated Milk and Enamel Caries in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Gunnel Svensater, Professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Malmö University
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Caries,Dental
Keywords: adolescents; flouridated milk; caries prevention; enamel caries; bitewing radiography
MeSH Terms: conditions — Dental Caries | interventions — Milk

STUDY DESIGN:
Intervention Model Description: Two parallel arms; an intervention group receiving doses of fluoride in water to add to milk and a control group receiving water to add to milk
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects and their parents/guardians, the clinicians performing the examinations, the staff-members delivering the packages with solutions to the subjects, the trial investigators and the outcome assessors were blind to the allocation and group assignment. The solutions were distributed to the subjects in tubes pre-labelled with code numbers. The tubes had the same design independent of the solution with fluoride or placebo.
  After the randomization, lists with code numbers were saved as sealed files in a safety-deposit box. The code was broken when the study was completed, and the assessment of the outcome measures were processed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The subjects in the intervention group received individually packaged daily doses of sodium fluoride solution in 0.5 ml sterile water to be added to 200 ml of milk
  Interventions: Dietary Supplement: sodium sodium fluoride solution (0.75 mg for subjects aged 12 and 1.0 mg for subjects aged 13)
- Control group (Placebo Comparator): Subjects in the control group received a daily dose of 0.5 ml sterile water to be added to 200 ml of milk.
  Interventions: Dietary Supplement: Subjects in the control group received a daily dose of 0.5 ml sterile water to be added to 200 ml of milk.

INTERVENTIONS:
Dietary Supplement: sodium sodium fluoride solution (0.75 mg for subjects aged 12 and 1.0 mg for subjects aged 13)
  Arms: Intervention
Dietary Supplement: Subjects in the control group received a daily dose of 0.5 ml sterile water to be added to 200 ml of milk.
  Arms: Control group

SUMMARY:
The goal of this trial is to investigate whether low daily doses of fluoridated milk, in addition to oral hygiene routines with fluoridated toothpaste, can prevent caries development in adolescents' teeth. The main questions it aims to answer are:

* Does fluoridated milk lower the number of caries lesions in teeth over time?
* Does fluoridated milk lower the number of enamel caries lesions over time? Researchers will compare an intervention group receiving doses of fluoride in water to add to milk and a control group receiving water to add to milk.

The 12-13 year participants will:

* be examined at a baseline and once yearly up to 2 years
* be provided directly with the doses every second month at their dental clinic
* take the fluid daily

DETAILED DESCRIPTION:
During the study, the participants were asked to continue with their usual oral hygiene regimes, including tooth-brushing twice a day with toothpaste containing fluorides as recommended by the Swedish National Board of Health and Welfare.

At their yearly visit to their dental clinic the participants were asked about their health status, use of antibiotics, lactose intolerance, daily consumption of milk, tooth brushing frequency, type of toothpaste and use of other fluoride additives. Information on adverse effects (dental pain, visit to other dental clinic, and antibiotics due to dental infection) was collected.

Caries registration was performed by visual-tactile and radiographic examinations at baseline and 1 and 2 years. Visual-tactile examination was performed by a dental practitioner under lighting with a mirror and occasionally with a probe. Caries status was classified for the occlusal/incisal, buccal and lingual surfaces and the proximal surfaces of incisors and cuspids according to the ICDAS criteria with code 0 (for sound), 1-3 (for enamel caries) and 4-6 (for dentine caries). ICDAS is an internationally applied system for caries detection used clinically (The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries (reference). Radiographic examination of the proximal surfaces of premolars and molars with one bitewing radiograph on each side of the mouth took place in the same session.

ELIGIBILITY:
Inclusion Criteria:

* adolescents of both sexes, aged 12-¬13
* healthy (no oral disease or systemic disease possibly affecting the oral cavity). Health declaration used in the dental clinic was utilized to confirm health status
* adolescents with permanent posterior teeth/no primary molar teeth present and second premolars in contact with the mesial surface of the first molars
* adolescents who, together with their parents or guardians, gave informed written consent to participate. Data confidentiality and the right to withdraw from the study at any time were warranted to the adolescents in writing.

Exclusion Criteria:

None

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Caries development in enamel and dentine | From enrollment to the end of intervention at 2 years
  caries increment measured as change/no change of DMFS (Decayed, Missing, Filled, Surfaces)

SECONDARY OUTCOMES:
Caries lesion arrest | From enrollment to the end of intervention at 2 years
  Number of caries lesions given the same ICDAS score at the visual examination of the smooth surfaces combined with number of caries lesions of the proximal surfaces given the same radiographic score at baseline and 2 years
Caries lesion progression | From enrollment to the end of intervention at 2 years
  Number of caries lesions given a higher ICDAS score at the visual examination of the smooth tooth surfaces combined with number of caries lesions of the proximal surfaces given a higher radiographic score at 2 years compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gunnel Svensäter, Principal Investigator — Malmö University
Locations (1):
- Faculty of Odontology, Malmo University, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Senneby A, Elfvin M, Stebring-Franzon C, Rohlin M. A novel classification system for assessment of approximal caries lesion progression in bitewing radiographs. Dentomaxillofac Radiol. 2016;45(5):20160039. doi: 10.1259/dmfr.20160039. Epub 2016 Apr 4. PMID 27043978
- [Derived] Rohlin M, Neilands J, Davies JR, Isberg PE, Wickstrom C, Svensater G. Fluoridated milk is effective in prevention of enamel caries in adolescents: a randomised trial. Acta Odontol Scand. 2025 Dec 29;84:673-684. doi: 10.2340/aos.v84.45271. PMID 41460820